CLINICAL TRIAL: NCT01854034
Title: Phase II Study of AUY922 in NSCLC Patients With Exon 20 Insertion Mutations in EGFR
Brief Title: Phase 2 Study of AUY922 in NSCLC Patients With Exon 20 Insertion Mutations in EGFR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-484
Record Dates: First submitted 2013-05-12; First posted 2013-05-15 (Estimated); Results first posted 2018-04-10 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Advanced disease; EGFR mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AUY922 Treatment Arm (Experimental): AUY922 administered once weekly via intravenous, 70 mg/m2
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — AUY922 administered intravenously once a week at 70mg/m2

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is being studied. It also means that the FDA has not yet approved the drug for your type of cancer or for any use outside of research studies.

It has been found that some people with NSCLC have a change (mutation) in a certain gene called the EGFR gene. This mutated gene helps cancer cells grow. The majority of NSCLC patients with EGFR mutations achieve good outcomes with erlotinib or other EGFR inhibitor therapies, with a high response rate, prolonged progression-free survival and possibly improved overall survival from therapy. However, the 4% of EGFR mutant patients that harbor an exon 20 insertion mutation historically have reaped little benefit from EGFR-directed therapy due to the low affinity of this mutation for direct EGFR inhibitors, especially erlotinib and gefitinib (see Yasuda et al, Lancet Oncol 2011). This group of patients is ideal for studying other targeted therapeutic strategies that could affect the oncogene mutation in EGFR via alternative mechanisms.

AUY922 is an investigational drug that may stop cancer cells from growing abnormally. This drug has been used in other research studies. Information from those other research studies suggests that AUY922 may be effective in killing cancer cells in patients with exon 20 insertion mutations in EGFR.

The purpose of this study is to test the safety of AUY922 and determine how well AUY922 works for participants with advanced NSCLC and exon 20 insertion mutations in EGFR.

DETAILED DESCRIPTION:
Interested patients will be asked to undergo some screening tests and procedures to confirm that they are eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that patients do not take part in the research study. If patients have had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures include: a medical history physical exam, performance status, assessment of tumor, EKG, electrocardiogram or multigated acquisition scan, eye exam, blood draw, blood pregnancy test, urine test and collection of a piece of the stored tumor tissue.

The study treatment is given in 21 day cycles. AUY922 is given by IV (into a vein). This is called an infusion. Patients will receive an infusion of AUY922 on days 1, 8 and 15 of each cycle (once per week). The infusion will take about 60 minutes.

A schedule of clinic visits for the study is summarized below.

Cycle 1, Day 1: physical exam, including measurement of vital signs and weight; performance status; EKG; blood draw; routine urine test Cycle 1, Day 2: EKG Cycle 1, Day 3: EKG Cycle 1, Day 8: Vital signs, performance status, EKG, questions about side effects and other medications taken Cycle 1, Day 15: Physical exam, including measurement of vital signs, performance status; EKG; blood draw; questions about side effects and other medications taken Note that in Cycle 1 patients will need to stay at (or return to) the clinic for the last EKG following the Day 1 AUY922 infusion, and come to the clinic on Days 2 and 3 for EKGs.

Cycle 2 and beyond, Day 1: physical exam, including measurement of vital signs and weight; performance status; EKG; blood draw; questions about side effects and other medications taken; routine urine test Cycle 2 and beyond, Day 8: Vital signs; performance status; EKG; questions about side effects and other medications taken Cycle 2 and beyond, Day 15: Physical exam, including measurement of vital signs; performance status; EKG; blood draw; questions about side effects and other medications taken.

Additional EKGs may be done at any time if the study doctor thinks it is necessary. A blood test to measure the amount of cardiac enzymes in the blood may be done whenever abnormal findings are suspected or seen on the EKG.

Additional tests and procedures:

* CT or MRI scans will be done to measure the disease about every 6 weeks.
* A blood pregnancy test, for women who can become pregnant, will be performed every 6 weeks or at any point in which pregnancy is suspected.
* A standard eye exam will be done on Cycle 3, Day 1. Additional eye exams will be done if patients experience any eye-related symptoms, such as changes in vision.

Within 1 week after the last dose of the study drug AUY922, patients will be asked to return to the clinic. At this visit the following will be done: physical examination, performance status, EKG, ECHO or MUGA scan, blood draw, urine test, eye exam, questions about side effects and other medications taken. Patients will be asked to return to the clinic a second time so investigators can follow-up on any ongoing side effects after stopping AUY922.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IV or recurrent NSCLC
* Measurable disease by RECIST 1.0
* Must have received at least one prior line of therapy for advanced lung cancer (no maximum number)
* Life expectancy of at least 12 weeks

Exclusion Criteria:

* Pregnant or breastfeeding
* Radiation within 2 weeks
* Cytotoxic chemotherapy or monoclonal antibodies within 4 weeks
* EGFR tyrosine kinase inhibitor within 2 weeks
* Other small molecule inhibitor within 2 weeks
* Experimental treatment within 30 days
* Prior treatment with any HSP90 or HDAC inhibitor compound
* Known and untreated brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AUY922
* Unresolved diarrhea greater than or equal to CTCAE version 4, grade 1
* Major surgery within 2 weeks of starting study drug or have not recovered from side effects of surgery
* Known disorders due to a deficiency in bilirubin glucuronidation
* Requiring use of therapeutic doses of warfarin (Coumadin)
* History of long QT syndrome
* History of clinically manifest ischemic heart disease, heart failure or left ventricular dysfunction
* Clinically significant ECG abnormalities
* Other clinically significant heart disease
* Currently receiving treatment with any medication which has a relative risk of prolonging the QTc interval or inducing Torsades de Pointes
* On a cardiac pacemaker
* Concurrent malignancies or invasive cancers diagnosed within 3 years except for adequately treated basal cell cancer of the skin or in situ cancer of the cervix
* Known to be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia Sequist, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Piotrowska Z, Costa DB, Oxnard GR, Huberman M, Gainor JF, Lennes IT, Muzikansky A, Shaw AT, Azzoli CG, Heist RS, Sequist LV. Activity of the Hsp90 inhibitor luminespib among non-small-cell lung cancers harboring EGFR exon 20 insertions. Ann Oncol. 2018 Oct 1;29(10):2092-2097. doi: 10.1093/annonc/mdy336. PMID 30351341

RESULTS

PARTICIPANT FLOW:
Groups:
- AUY922 Treatment Arm: AUY922 administered intravenously once a week at 70mg/m2
Period: Overall Study
Arm/Group | AUY922 Treatment Arm
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AUY922 Treatment Arm
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 60 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29
Median Prior Lines of Therapy [Median (Full Range); unit: Therapies] | 1 [1 to 5]
Number of Participants with prior EGFR TKI [Count of Participants; unit: Participants] — epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor (TKI)
  Participants | 6
Baseline ECOG PS [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
  * 0: Asymptomatic (Fully active, able to carry on all pre-disease activities without restriction)
  * 1: Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
  * 2: Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
  Participants
    0 | 9
    1 | 18
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The number of participants that achieved a response to treatment as assessed by Response Evaluation Criteria is Solid Tumors (RECIST). Response is defined as having achieved either a complete response (CR) or a partial response (PR).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the start of treatment until the time of disease progression, median duration of follow-up of about 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922 Treatment Arm
Number analyzed (Participants) | 29
Participants | 5

2. Secondary Outcome: Median Progression Free and Overall Survival
Description: Overall survival (OS) is measured from the start of treatment until the time of death. Progression free survival is measured from the start of treatment until the time of death or disease progression as assessed by RECIST. Progressive disease is defined as having at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study with at least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions denotes disease progression.
Time Frame: From the start of treatment until the time or death or disease progression
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AUY922 Treatment Arm
Number analyzed (Participants) | 29
Months
  Overall Survival | 9.9 [4.5 to 19.2]
  Progression Free Survival | 2.8 [1.3 to 5.6]

3. Secondary Outcome: The Number of Participants With Treatment Related Serious Adverse Events
Description: The number of participants with serious adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) that were deemed to be possibly, probably, or definitely related to study treatment as determined by the treating physician.
Time Frame: From the start of treatment until 28 days after the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | AUY922 Treatment Arm
Number analyzed (Participants) | 29
Participants | 6

4. Secondary Outcome: Exon 20 EGFR Mutations Among Participants That Responded to Treatment
Description: The specific exon 20 epidermal growth factor receptor (EGFR) mutations among participants that achieved either a partial response or complete response as assessed by RECIST. The EGFR mutations were assessed from biopsies taken at baseline and then the baseline mutations were categorized by disease response.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to < 10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline, at the time of response
Measure: Number; unit: participants
Arm/Group | AUY922 Treatment Arm
Number analyzed (Participants) | 5
participants
  Complete Response : D770_P772dup | 1
  Partial Response : N771insGF | 1
  Partial Response : D770_N771insSVD | 1
  Partial Response : P772_H773dupPH | 1
  Partial Response : P773dup | 1

ADVERSE EVENTS:
Time Frame: From baseline until 28 days after the last dose of the study drug was received (±7 days). Treatment is continued until: > Disease progression. > Intercurrent illness that prevents further administration of treatment, > Unacceptable adverse event(s), > Participant decides to withdraw from the study, or > General or specific changes in the participant's condition render the participant unacceptable for further treatment in the opinion of the treating investigator
Description: Serious adverse events are defined as grade 3 or higher adverse events deemed to at least possibly related to the study drug.
Arm/Group | AUY922 Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 6/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUY922 Treatment Arm (N=29)
Eye Disorder- Other (Eye disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUY922 Treatment Arm (N=29)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Alanine aminotransferase increased (Investigations) | 2 (2)
Allergic reaction (Immune system disorders) | 4 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Anxiety (Psychiatric disorders) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Blurred vision (Eye disorders) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (10)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cataract (Eye disorders) | 2 (3)
Cholesterol high (Investigations) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 23 (30)
Dizziness (Nervous system disorders) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Edema limbs (General disorders) | 4 (4)
Eye disorders - Other, specify (Eye disorders) | 21 (33)
Fatigue (General disorders) | 23 (35)
Fever (General disorders) | 2 (2)
Flashing lights (Eye disorders) | 3 (3)
Floaters (Eye disorders) | 4 (4)
Gait disturbance (General disorders) | 4 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 5 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 12 (16)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 11 (23)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (14)
Hypothyroidism (Endocrine disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 5 (5)
Insomnia (Psychiatric disorders) | 7 (7)
Musculoskeletal and connective tissue disorders - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (4)
Night blindness (Eye disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 6 (6)
Pain (General disorders) | 11 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 4 (4)
Thromboembolic event (Vascular disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (5)
Weight loss (Investigations) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT01854034/Prot_SAP_000.pdf